CLINICAL TRIAL: NCT01914783
Title: Experimental Exposure to Air Pollutants and Sympathetic Nerve Activity in Human Subjects
Acronym: Particles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Collaborators: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Responsible Party: Principal Investigator, Prof. Dr. Jens Jordan, Professor Dr. med. Jens Jordan, Hannover Medical School
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MHH-Particles EK-6142
Record Dates: First submitted 2013-07-30; First posted 2013-08-02 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Cardiovascular Morbidity
Keywords: air pollution; ozone; fine particle; cytokine; chemokine; oxidative stress; inflammation; heart rate variability; autonomic nervous system; sympathetic nerve activity; plasma catecholamine
MeSH Terms: conditions — Inflammation | interventions — Particulate Matter; Ozone; Environment, Controlled

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ultrafine particles (Experimental): Subjects will be exposed to ultrafine particles for three hours in an exposure chamber. During that time participants will perform intermittent bicycle ergometer training. Training intensity is adjusted individually to increase ventilation to 20 l/min/m². During exposure, heart rate will be monitored continuously via ECG. Blood pressure will be measured every 15 minutes. Ultrafine elemental carbon black particles are generated using a commercially available electric spark generator. Particle number, mass, and size distribution will be monitored during exposure.
  Interventions: Other: ultrafine particles
- ultrafine particles and ozone (Active Comparator): Subjects will be exposed to ultrafine particles for three hours in an exposure chamber. During that time participants will perform intermittent bicycle ergometer training. Training intensity is adjusted individually to increase ventilation to 20 l/min/m². During exposure, heart rate will be monitored continuously via ECG. Blood pressure will be measured every 15 minutes. Ultrafine elemental carbon black particles are generated using a commercially available electric spark generator. Particle number, mass, and size distribution will be monitored during exposure.Ozone is generated from medical oxygen in order to maintain a concentration of 250 ppb.
  Interventions: Other: ultrafine particles and ozone
- clean air (Placebo Comparator): Subjects will be exposed to clean air for three hours in an exposure chamber controlled for temperature, humidity, and gas/particle composition. During that time they will perform intermittent bicycle ergometer training for 15 minutes alternating with 15 minutes rest. Training intensity is adjusted individually to increase ventilation to 20 l/min/m². During exposure, heart rate will be monitored continuously via ECG. The blood pressure will be measured in time intervals of 15 minutes.
  Interventions: Other: clean air

INTERVENTIONS:
Other: ultrafine particles — exposure to ultrafine particles
  Arms: ultrafine particles
Other: ultrafine particles and ozone — exposure to ultrafine particles and ozone
  Arms: ultrafine particles and ozone
Other: clean air — Exposure to clean air.
  Arms: clean air

SUMMARY:
The primary hypothesis of the study is that in healthy elderly subjects experimental exposure to air pollutants increases sympathetic nervous system activity compared with sham (clean air) exposure. The secondary hypothesis of the study is that combined experimental exposure to air pollutants (particles + ozone) increases sympathetic nervous system activity to a greater extent than does the exposure to particles alone.

DETAILED DESCRIPTION:
In a randomized, double-blind, and cross-over fashion, the participants will be exposed to clean air, ultrafine particles, or ultrafine particles and ozone in an exposure chamber. The investigators will determine blood pressure, heart rate, respiration as well as cardiac output and directly record sympathetic vasomotor tone using the microneurography technique. To elucidate the underlying mechanisms through which particles and ozone affect the autonomic nervous system, the investigators will assess the local and systemic inflammatory response as well as the changes in neurotrophic factors in sputum and blood. In addition, the activation of inflammatory cells in sputum and blood will be analyzed at different points in time after exposures. Changes in sympathetic activity will be correlated with the degree of airway inflammation and oxidative stress assessed in induced sputum and blood. This study will provide important insight in the mechanisms through which air pollution, particularly ultrafine particle exposure, increases cardiovascular risk in human subjects and generate a human model for mechanistic and therapeutic studies.

ELIGIBILITY:
Inclusion Criteria:

* Elderly man or postmenopausal woman older than 50 years of age.
* Signed written informed consent.

Exclusion Criteria:

* Smoker.
* Cardiovascular and/or pulmonary disease.
* Medication with relevant impact on autonomic system function, e. g. norepinephrine reuptake inhibitors. Stable medication with slight to moderate autonomic effects is tolerable.
* Subject is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol.
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
* Subject unlikely to comply with protocol, e. g. uncooperative attitude or unlikelihood of completing the study.
* Known hypersensitivity to ozone.
* History of drug or alcohol abuse. Particles Study - Protocol version: October 19, 2012 14
* Blood donation of more than 500 mL during the previous 3 months.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Muscle sympathetic nerve activity (MSNA) | 2.5 hours after exposure to clean air, to ultrafine particles, or to a combination of ultrafine particles and ozone
  Change of sympathetic vasoconstrictor nerve activity directed to skeletal muscle expressed as sympathetic bursts per minute. The primary hypothesis of the study is that in healthy elderly subjects experimental exposure to air pollutants increases sympathetic nervous system activity compared with sham (clean air) exposure.

SECONDARY OUTCOMES:
MSNA burst incidence | 2.5 hours after exposure to clean air, to ultrafine particles, or to a combination of ultrafine particles and ozone
  Change of MSNA expressed as bursts/100 heart beats.
total MSNA | 2.5 hours after exposure to clean air, to ultrafine particles, or to a combination of ultrafine particles and ozone
  Change of MSNA expressed as burst area/min.

OTHER OUTCOMES:
Blood pressure | 2.5 hours after exposure to clean air, to ultrafine particles, or to a combination of ultrafine particles and ozone
  Change of blood pressure in mmHg.
Heart rate | 2.5 hours after exposure to clean air, to ultrafine particles, or to a combination of ultrafine particles and ozone
  Change of heart rate in beat per minute.
Cardiac output | 2.5 hours after exposure to clean air, to ultrafine particles, or to a combination of ultrafine particles and ozone
  Change of cardiac output in l/min.
Total peripheral resistance | 2.5 hours after exposure to clean air, to ultrafine particles, or to a combination of ultrafine particles and ozone
  Change in total peripheral resistance expressed as dyn*s/cm^5.
Heart rate variability. | 2.5 hours after exposure to clean air, to ultrafine particles, or to a combination of ultrafine particles and ozone
  Change in heart rate variability parameters in the time and frequency domain.
Plasma norepinephrine concentration | 2.5 hours after exposure to clean air, to ultrafine particles, or to a combination of ultrafine particles and ozone
  Change of plasma norepinephrine in ng/l.
Plasma renin concentration | 2.5 hours after exposure to clean air, to ultrafine particles, or to a combination of ultrafine particles and ozone
  Change of plasma renin concentration in
Baroreflex sensitivity | 2.5 hours after exposure to clean air, to ultrafine particles, or to a combination of ultrafine particles and ozone
  Change in baroreflex sensitivity expressed as ms/mmHg.
Inflammation parameters | 3.5 hours after exposure to clean air, to ultrafine particles, or to a combination of ultrafine particles and ozone
  Change of the percentage of neutrophils in induced sputum.
Oxidative stress parameters | 2.5 hours after exposure to clean air, to ultrafine particles, or to a combination of ultrafine particles and ozone
  Change of plasma malondialdehyde(MDA)concentration.
Correlation between inflammation, oxidative stress and cardiovascular regulation | 2.5 hours after exposure to clean air, to ultrafine particles, or to a combination of ultrafine particles and ozone
  Correlation coefficients between changes in parameters for inflammation and oxidative stress with changes in cardiovascular parameters.
Forced expiratory volume in one second (FEV1) | 2.5 hours after exposure to clean air, to ultrafine particles, or to a combination of ultrafine particles and ozone
  Change in FEV1 in l
Forced vital capacity (FVC) | 2.5 hours after exposure to clean air, to ultrafine particles, or to a combination of ultrafine particles and ozone
  Change in FVC in l.
Percentage of neutrophils in peripheral blood | 2.5 hours after exposure to clean air, to ultrafine particles, or to a combination of ultrafine particles and ozone
  Change of percentage of neutrophils in peripheral blood.

CONTACTS AND LOCATIONS:
Locations (1):
- Hannover Medical School, Hanover, Germany

REFERENCES:
- [Background] Tank J, Biller H, Heusser K, Holz O, Diedrich A, Framke T, Koch A, Grosshennig A, Koch W, Krug N, Jordan J, Hohlfeld JM. Effect of acute ozone induced airway inflammation on human sympathetic nerve traffic: a randomized, placebo controlled, crossover study. PLoS One. 2011 Apr 8;6(4):e18737. doi: 10.1371/journal.pone.0018737. PMID 21494635